CLINICAL TRIAL: NCT01236716
Title: A Randomized Phase II Clinical Trial of Nab-Paclitaxel and Carboplatin Compared With Gemcitabine and Carboplatin as First-line Therapy in Advanced Squamous Cell Carcinoma of Lung
Brief Title: Nab-Paclitaxel Treatment in Advanced Squamous Cell Carcinoma of Lung
Acronym: C-TONG1002
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Society of Lung Cancer (Other)
Responsible Party: Principal Investigator, Yi-Long Wu, Professor, Chinese Society of Lung Cancer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-TONG1002
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: squamous cell carcinoma of lung; Albumin bound paclitaxel; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Albumin paclitaxel plus carboplatin (Experimental): Treatment of Albumin paclitaxel plus carboplatin
  Interventions: Drug: Albumin paclitaxel plus carboplatin
- Gemcitabine plus carboplatin (Active Comparator): Treatment of Gemcitabine plus carboplatin
  Interventions: Drug: Gemcitabine plus carboplatin

INTERVENTIONS:
Drug: Albumin paclitaxel plus carboplatin — Patients receive carboplatin AUC=5 q3w and nab-p 135 mg/m2 weekly for 2 weeks (on days 1 and 8 of a 21-day cycle), followed by a week of rest.
  Other Names: Abraxane(Albumin-bound paclitaxel,nab-P)
  Arms: Albumin paclitaxel plus carboplatin
Drug: Gemcitabine plus carboplatin — Patients receive carboplatin AUC=5 q3w and gemcitabine 1250 mg/m2 weekly for 2 weeks (on days 1 and 8 of a 21-day cycle), followed by a week of rest.
  Other Names: Gemzar(Gemcitabine)
  Arms: Gemcitabine plus carboplatin

SUMMARY:
This trial is to study the efficacy of nab-PC vs. GC and evaluate toxicity of nab-PC in advanced squamous cell cancer of lung. The correlation between the efficacy of nab-PC and some biomarkers is also to be evaluated.

DETAILED DESCRIPTION:
Albumin-bound paclitaxel(nab-P) utilizes the albumin binding proteins,such as (gp60)/caveolin-1 (CAV1) and SPARC(secreted protein acidic and rich in cysteine), achieving high intratumoral paclitaxel accumulation. It is reported that CAV1 is overexpressed in squamous cell cancer(SQC), so it is possible that nab-PC is more highly active than GC in SQC of lung.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, histological documented stage IIIB (not amenable for radical regional therapy) or stage IV squamous cell carcinoma of lung. At least one measurable lesion as defined by RECIST criteria.
* At least 18 years of age.
* ECOG PS 0~1
* Patients have no previously malignant tumor history except cured cervical carcinoma in situ, basal cell carcinoma or superficial bladder cancer. Patients are also eligible if they have received a chemotherapy regimen as neoadjuvant or adjuvant chemotherapy and the disease recurred over 12 months since the finishing of neoadjuvant or adjuvant chemotherapy.
* neutrophil ≥ 1.5 x 109 /L, Hemoglobin > 90 g/L, Platelet count > 100x109/L.
* Total bilirubin ≤ 1.5 x upper limit of normal. ALT and AST < 2.5 x upper limit of normal without liver metastasis, ALT and AST < 5 x upper limit of normal with liver metastasis. Serum creatinine < 1.5 x upper limit of normal.
* Urine pregnancy test is negative for woman.
* Estimated life expectancy is at least 3 months.
* Patient comply with the clinical trial protocal.
* Informed consent must be signed.

Exclusion Criteria:

* Patients who are currently undergoing other anti-tumor therapy.
* Patients who was enrolled in any other clinical trial within 4 weeks of study entry.
* Any physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of any study medication or render the subject at high risk from treatment.
* Central nervous system (CNS) tumor or metastatic tumor.
* Serious mental disorder.
* Serious dysgnosia.
* Other serious comorbidity.
* Alcohol or drug dependence.
* Previously allergic to drugs used in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2010-11; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Overall response rate(ORR) | 18weeks
  ORR is evaluated after at most 6 cycles of chemotherapy, which may cost 18 weeks.

SECONDARY OUTCOMES:
Response duration, progression free survival, overall survival, safety profile | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Wu Yilong, professor, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Wang Z, Huang C, Yang JJ, Song Y, Cheng Y, Chen GY, Yan HH, Ben XS, Wang BC, Xu CR, Jiang BY, Zhou Q, Chen HJ, Wu YL. A randomised phase II clinical trial of nab-paclitaxel and carboplatin compared with gemcitabine and carboplatin as first-line therapy in advanced squamous cell lung carcinoma (C-TONG1002). Eur J Cancer. 2019 Mar;109:183-191. doi: 10.1016/j.ejca.2019.01.007. Epub 2019 Feb 7. PMID 30739019
- [Derived] Yang JJ, Huang C, Chen GY, Song Y, Cheng Y, Yan HH, Zhou Q, Wu YL. A randomized phase II clinical trial of nab-paclitaxel and carboplatin compared with gemcitabine and carboplatin as first-line therapy in locally advanced or metastatic squamous cell carcinoma of lung. BMC Cancer. 2014 Sep 20;14:684. doi: 10.1186/1471-2407-14-684. PMID 25239521
- [Derived] Gold KA, Wistuba II, Kim ES. New strategies in squamous cell carcinoma of the lung: identification of tumor drivers to personalize therapy. Clin Cancer Res. 2012 Jun 1;18(11):3002-7. doi: 10.1158/1078-0432.CCR-11-2055. Epub 2012 Mar 29. PMID 22461458